CLINICAL TRIAL: NCT04274257
Title: Double-Blind, Parallel-group Comparison, Investigators Initiated Phase II Clinical Trial of IDEC-C2B8 (Rituximab) in Patients With Systemic Sclerosis
Brief Title: A Study of the Efficacy and Safety of Rituximab in Participants With Systemic Sclerosis
Acronym: DesiReS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tokyo University (Other)
Collaborators: Japan Agency for Medical Research and Development (Other Government); Zenyaku Kogyo Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ayumi Yoshizaki, Principal Investigator, Tokyo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017019-11DX
Record Dates: First submitted 2020-02-13; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Scleroderma, Systemic; Skin Sclerosis; Lung Fibrosis; Autoimmune Diseases; Collagen Diseases
MeSH Terms: conditions — Scleroderma, Systemic; Pulmonary Fibrosis; Autoimmune Diseases; Collagen Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Double-Blind Placebo (Placebo Comparator): Participants will receive double-blind matching placebo from baseline until week 24. Participants may then receive open-label rituximab from weeks 24 to 48.
  Interventions: Drug: Double-Blind Placebo
- Double-Blind Rituximab (Experimental): Participants will receive double-blind rituximab from baseline until week 24. Participants may then receive open-label rituximab from weeks 24 to 48.
  Interventions: Drug: Double-Blind Rituximab

INTERVENTIONS:
Drug: Double-Blind Placebo — The 4-week treatment period (four 375 mg/m2 doses at 1-week intervals) and subsequent 20-week follow-up period constitute one cycle of treatment.
  In the double-blind period, one cycle of placebo will be administered. In the active drug period, one additional cycle (rituximab) will be administered.
  Arms: Double-Blind Placebo
Drug: Double-Blind Rituximab — The 4-week treatment period (four 375 mg/m2 doses at 1-week intervals) and subsequent 20-week follow-up period constitute one cycle of treatment.
  In the double-blind period, one cycle of rituximab will be administered. In the active drug period, one additional cycle (rituximab) will be administered.
  Arms: Double-Blind Rituximab

SUMMARY:
This study evaluates the efficacy and safety of rituximab compared with placebo in SSc patients. This study consists of a 24-week, double-blind, placebo-controlled period followed by a 24-week active drug treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfill the diagnostic criteria for systemic sclerosis defined in the 2016 edition of the Clinical Practice Guidelines for Systemic Sclerosis and have an mRTSS of 2 (moderate) or higher for skin sclerosis
2. Aged 20 or older and younger than 80 at the time of consent
3. Have an expected survival of at least 6 months (and expected to allow 6 months of observation)
4. Fulfill the following criteria related to concomitant medications/therapies:

   * Not received corticosteroids equivalent to more than 10 mg/day of prednisolone within 2 weeks before the start of study treatment; and
   * Not received antifibrotic agents (like nintedanib, pirfenidone, tocilizumab), other investigational products, immunosuppressants (cyclophosphamide, mycophenolate mofetil, ciclosporin, tacrolimus, azathioprine, and mizoribine), high-dose intravenous immunoglobulin, or imatinib 4 weeks prior to the start of study treatment.
5. Provided written consent to participate in the study

Exclusion Criteria:

1. Present with pulmonary hypertension* associated with systemic sclerosis

   *: The patient will undergo echocardiography during the pre-treatment observation period to exclude pulmonary hypertension. The patient will be required to undergo examination by an expert (eg, at the Department of Cardiovascular Medicine) if systolic pulmonary artery pressure exceeds 35 mmHg.
2. Have serious complications (eg, renal crisis) associated with systemic sclerosis (excluding interstitial pneumonia**)

   **: Patients with interstitial pneumonia will be excluded if the criterion 3) below is met.
3. Have only poor respiratory reserve (%VC or %DLco, both calculated using the "estimation equation more suitable for Japanese," is less than 60% or 40%, respectively)
4. Known to have HIV antibodies
5. Have a positive result for any of the following: HBs antigen, HBs antibody, HBc antibody, and HCV antibody (this criterion does not apply to a positive test for hepatitis B clearly attributable to hepatitis vaccination)
6. Have serious bacterial/fungal infections
7. Have a serious liver disease (AST [GOT] or ALT[GPT] of ≥ 300 IU)
8. Have a serious renal disease (serum creatinine ≥ 2.0 mg/dL)
9. Have severe heart disease
10. Have active tuberculosis
11. Have any known malignancy or a history of malignancy within the past 5 years
12. Have a history of serious infections
13. Have a history of serious hypersensitivity or anaphylactic reactions to any component of rituximab or to mouse proteins
14. Pregnant, postpartum, and lactating women
15. Refuse to practice contraception from the time of consent to at least 12 months after study completion
16. Have any disease or physical/psychiatric conditions that make study participation difficult/inappropriate
17. Received other investigational products within 12 weeks prior to the study treatment or are participating in other clinical research/studies
18. Smoked within 12 weeks prior to the date of consent
19. Is determined by the investigator (or sub-investigator) to be ineligible for the study for any other reason

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Change in Modified Rodnan Total Skin Thickness Score (mRTSS) during double-blind period | From baseline to week 24
  Absolute change from pre-treatment observation period in skin sclerosis at week 24 of treatment in the double-blind phase, assessed by mRTSS. mRTSS ranging from 0 (normal) to 3 (severe skin thickening) across 17 different body parts. The total score is the sum of the individual skin scores for all these sites, and ranges from 0 to 51 units.

SECONDARY OUTCOMES:
Change in percent FVC measured in respiratory function test | From baseline to week 24
Change in percent DLco measured in respiratory function test | From baseline to week 24
Change in TLC measured in respiratory function test | From baseline to week 24
Change in serum levels of KL-6 | From baseline to week 24
Change in serum levels of SP-D | From baseline to week 24
Change in serum levels of SP-A | From baseline to week 24
Change in percentage of interstitial shadow in lungs by high-resolution computed tomography | From baseline to week 24
Change in skin thickness measured following biopsy specimen | From baseline to week 24
Change in HRQOL index measured using MOS 36 Item Short-Form Health Survey | From baseline to week 24
Change in QOL index of SSc patients, assessed using the Health Assessment Questionnaire Disability Index (HAQ-DI) | From baseline to week 24
Change in serum antinuclear antibody titers | From baseline to week 24
Change in serum levels of anti-centromere antibodies | From baseline to week 24
Change in serum levels of anti-Scl-70 antibodies | From baseline to week 24
Change in serum levels of anti-RNA polymerase III antibodies | From baseline to week 24
Change in serum levels of anti-ssDNA antibodies | From baseline to week 24
Change in serum levels of anti-dsDNA antibodies | From baseline to week 24
Change in serum levels of anti-CL antibodies | From baseline to week 24
Change in serum levels of anti-β2-GP1 antibodies | From baseline to week 24
Change in serum levels of lupus anticoagulant | From baseline to week 24
Change in serum levels of anti-SS-A antibodies | From baseline to week 24
Change in serum levels of anti-SS-B antibodies | From baseline to week 24
Change in serum levels of anti-cANCA | From baseline to week 24
Change in serum levels of anti-p-ANCA | From baseline to week 24
Change in serum levels of anti-U1-RNP antibodies | From baseline to week 24
Change in serum levels of IgG | From baseline to week 24
Change in serum levels of IgM | From baseline to week 24
Change in serum levels of IgA | From baseline to week 24
Change in blood CD19+ B cell count | From baseline to week 24
Change in blood CD20+ B cell count | From baseline to week 24
Change in blood CD3+ T cell count | From baseline to week 24
Expression of human anti-rituximab antibodies | From baseline to week 24
Overall incidence, severity, causal relationship, and outcome of adverse events | From baseline to week 48
Incidence of rituximab infusion reactions | From baseline to week 48
PK profile of rituximab: Area under concentration-time curve from time 0 to final observation (AUC0-t) | From baseline to week 48
PK profile of rituximab: maximum serum concentration after dosing (Cmax) | From baseline to week 48
PK profile of rituximab: time to maximum concentration (tmax) | From baseline to week 48
PK profile of rituximab: terminal half-life (t1/2) | From baseline to week 48
PK profile of rituximab: mean residence time | From baseline to week 48
PK profile of rituximab: clearance | From baseline to week 48
PK profile of rituximab: volume of distribution | From baseline to week 48

CONTACTS AND LOCATIONS:
Overall Officials: Ayumi Yoshizaki, MD, PhD, Principal Investigator — Tokyo University
Locations (4):
- Japan (4):
  - University of Fukui Hospital, Fukui
  - Chukyo Hospital, Nagoya
  - The University of Tokyo Hospital, Tokyo
  - University of Tsukuba Hospital, Tsukuba

REFERENCES:
- [Derived] Ebata S, Yoshizaki A, Oba K, Kashiwabara K, Ueda K, Uemura Y, Watadani T, Fukasawa T, Miura S, Yoshizaki-Ogawa A, Okiyama N, Kodera M, Hasegawa M, Sato S. Safety and efficacy of rituximab in systemic sclerosis (DESIRES): open-label extension of a double-blind, investigators-initiated, randomised, placebo-controlled trial. Lancet Rheumatol. 2022 Aug;4(8):e546-e555. doi: 10.1016/S2665-9913(22)00131-X. Epub 2022 Jun 28. PMID 38294008
- [Derived] Ebata S, Yoshizaki A, Oba K, Kashiwabara K, Ueda K, Uemura Y, Watadani T, Fukasawa T, Miura S, Yoshizaki-Ogawa A, Asano Y, Okiyama N, Kodera M, Hasegawa M, Sato S. Safety and efficacy of rituximab in systemic sclerosis (DESIRES): a double-blind, investigator-initiated, randomised, placebo-controlled trial. Lancet Rheumatol. 2021 Jul;3(7):e489-e497. doi: 10.1016/S2665-9913(21)00107-7. Epub 2021 May 26. PMID 38279402
- [Derived] Ebata S, Oba K, Kashiwabara K, Ueda K, Uemura Y, Watadani T, Fukasawa T, Miura S, Yoshizaki-Ogawa A, Yoshihide A, Yoshizaki A, Sato S. Predictors of rituximab effect on modified Rodnan skin score in systemic sclerosis: a machine-learning analysis of the DesiReS trial. Rheumatology (Oxford). 2022 Nov 2;61(11):4364-4373. doi: 10.1093/rheumatology/keac023. PMID 35136981